CLINICAL TRIAL: NCT04529941
Title: Using Electrical Nerve Stimulation to Control Atrial Fibrillation
Acronym: STALL-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Indiana University (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Peng-Sheng Chen, Staff Physician, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00000581; 7OT2OD028190-02 (NIH)
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Results first posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Equipment and Supplies

STUDY DESIGN:
Intervention Model Description: Patients will have a 1:1 randomization to receive subcutaneous electrical nerve stimulation (ScNS) to observe if the stimulation can reduce atrial fibrillation burden in patients with symptomatic atrial fibrillation (AF). All subjects will undergo the implant of a neurostimulator lead.
  The experimental group will receive stimulation and the control group will not receive stimulation. All subjects will complete the same follow up visits comparing the 2 groups. The control group will have an option to cross over to the experimental group 3 weeks post-randomization to receive the stimulation. They will repeat the baseline visit, procedure visit and all follow-up visits post-procedure.
Who Masked: Participant
Masking Description: Subjects will not be aware whether the ScNS is turned on or off. However, after three weeks from the initial surgery, control subjects that decide to the second procedure will be aware of what group they were randomized to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Experimental Group (Experimental): Will receive stimulation ScNS at 3.5mA output
  Interventions: Device: Device Implant with Active Treatment
- Control Group (Sham Comparator): Does not receive therapy
  Interventions: Device: Device Implant without Active Treatment

INTERVENTIONS:
Device: Device Implant with Active Treatment — ScNS at 3.5mA output for 2 weeks
  Arms: Experimental Group
Device: Device Implant without Active Treatment — No device output for 2 weeks
  Arms: Control Group

SUMMARY:
The purpose of this study is to examine if sending mild electrical signals just under your skin will improve atrial fibrillation symptoms by controlling your heart rate.

DETAILED DESCRIPTION:
Patients will have a 1:1 randomization to receive subcutaneous electrical nerve stimulation (ScNS) to observe if the stimulation can reduce atrial fibrillation burden in patients with symptomatic atrial fibrillation (AF). All subjects will undergo the implant of a neurostimulator lead. The experimental group will receive stimulation and the control group will not receive stimulation. All subjects will complete the same follow up visits to compare the 2 groups.

Primary Objective: To test the hypothesis that chronic subcutaneous nerve stimulation can reduce AF burden in patients with severe symptomatic AF unresponsive to conventional therapies

The secondary objective:

To test the hypotheses that the effect of ScNS on the following endpoints is different between the two randomization groups:

1. Time-dependent reduction of AF burden
2. Effects of ScNS on ventricular rate control during AF
3. Reduction of SKNA
4. Improvement of quality of life

The study will enroll patients with symptomatic atrial fibrillation unresponsive to conventional therapy defined by not responding to at least 1 antiarrhythmic drug. The study will enroll 30 patients, including 15 men and 15 women between the 18 and 75 years old. There will be no sex/gender/racial/ethnic based exclusion. Patients will be enrolled from the Cedars Sinai Medical Center.

The patients will undergo surgical implantation of an externalized lead under the skin on the chest wall. The wire is then connected to a neurostimulator. The experimental group (Group A) will receive ScNS (3.5mA) for two weeks. The sham group (Group B) will receive sham (0 mA) stimulation for two weeks. The AF burden will be assessed by a 7-day mobile cardiac telemetry device provided by Preventice. An additional mobile cardiac telemetry device, Bittium Faros, will also be worn at similar time points to monitor skin sympathetic nerve activity. An Apple watch will be used to collect additional information on the frequencies of AF between the Baseline Visit until the 3 Month Visit 7 Day Mobile Cardiac Telemetry is complete. After completion of the week 3 visit, the sham group (Group B) will be able to receive ScNS (3.5 mA) for two weeks. The AF burden will be assessed post-procedure by mobile cardiac telemetry by Preventice and Bittium Faros

Study duration: 36 Months

Subject duration: up to 5 months.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years of age
* Symptomatic Paroxysmal AF.

  * Symptomatic paroxysmal AF is defined by AF with patient-reported perception of one or more of the following symptoms: palpitations, dizziness/presyncope, syncope, dyspnea, chest pain, malaise, and fatigue and activity intolerance.
  * There is at least one ECG-documented AF episode.
* Unresponsive to conventional therapy is defined by not responding to at least 1 antiarrhythmic drug (class I, class III, or atrioventricular nodal blocker).
* The left atrial size <50 mm by transthoracic echocardiography documented by eligibility visit echocardiogram
* Documented atrial fibrillation as defined as atrial fibrillation >30 seconds in duration with an atrial fibrillation burden determined by a minimum of 7 days of continuous ePatch monitoring within 6 months before surgery.

Exclusion Criteria:

* Patients without AF episodes during monitoring period will be excluded from the study and count as screen failure
* Left ventricular ejection fraction <40%
* Heart failure with functional classes III or IV
* Recurrent vasovagal syncope
* Valvular AF (severe mitral regurgitation, mitral stenosis)
* Congenital heart diseases
* Wolff Parkinson-White Syndrome
* Stroke within the past 6 months
* Any history of myocardial infarction
* Malignancies with a life expectancy of < 1 year
* A history of ablation procedures to treat left atrial tachyarrhythmias or other serious comorbidity
* Any history of sustained ventricular tachycardia (VT) defined by (1) > 30 s in duration or (2) < 30 s in duration, but is associated with hemodynamic consequences such as hypotension and syncope.
* Patients with a vagal nerve stimulator
* Active thyrotoxicosis
* Sick sinus syndrome with symptomatic bradycardia
* Heart rate < 50 beats per minute in sinus rhythm on 12-lead ECG
* Systolic blood pressure < 90 mm Hg
* Any experimental medication concomitantly or within 4 weeks of participation in the study
* Subjects with cardiac implantable electronic device (CIED) such as pacemakers and implantable cardioverter-defibrillators (ICDs)
* Pre-existing neuromodulation devices, such as vagal nerve stimulators, spinal cord stimulators and sacral nerve stimulators
* People with a history of allergy to ECG electrodes, adhesive tape, or nylon
* Pregnant women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2024-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peng-Sheng Chen, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- CedarsSinaiMC, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 46 subjects were enrolled in the study and underwent mobile cardiac telemetry and echocardiogram to determine eligibility. Out of this group, 16 subjects were deemed eligible and completed a baseline visit prior to the procedure and randomization.
Groups:
- Control (Sham) Group: Does not receive therapy
  Device Implant without Active Treatment: No device output for 2 weeks.
  After Week 3, has the option to forego the Week 12 Follow Up visit and, instead, repeat device implantation to crossover to the experimental group to receive stimulation. Will repeat all visits and assessments.
Period: Device Implantation and Randomization
Arm/Group | Experimental Group | Control (Sham) Group
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Week 1 Follow Up
Arm/Group | Experimental Group | Control (Sham) Group
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Week 2 Follow Up and Device Removal
Arm/Group | Experimental Group | Control (Sham) Group
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Week 3 Follow Up
Arm/Group | Experimental Group | Control (Sham) Group
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Crossover Option
Arm/Group | Experimental Group | Control (Sham) Group
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0
Period: Week 12/Month 3 Follow Up
Arm/Group | Experimental Group | Control (Sham) Group
Started | 8 | 7
Completed | 7 | 7
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Due to low baseline burden (<1%), 2 randomized subjects from each group were excluded from efficacy analysis. Therefore, although randomized, baseline measures were not and analyzed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Group | Control Group | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Due to low baseline burden (<1%), 2 randomized subjects from each group were excluded from efficacy analysis.
  years | 64.0 (7.4) | 57.8 (12.3) | 60.9 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Due to low baseline burden (<1%), 2 randomized subjects from each group were excluded from efficacy analysis.
  Participants
    Female | 3 | 1 | 4
    Male | 3 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Due to low baseline burden (<1%), 2 randomized subjects from each group were excluded from efficacy analysis.
  Participants
    Hispanic or Latino | 0 | 0 | 0
    Not Hispanic or Latino | 6 | 6 | 12
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Due to low baseline burden (<1%), 2 randomized subjects from each group were excluded from efficacy analysis.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 1 | 1 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 1 | 1 | 2
    White | 4 | 4 | 8
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Population: Due to low baseline burden (<1%), 2 randomized subjects from each group were excluded from efficacy analysis.
  participants
    United States | 6 | 6 | 12
Smoking [Count of Participants; unit: Participants] — Population: Due to low baseline burden (<1%), 2 randomized subjects from each group were excluded from efficacy analysis.
  Participants
    None | 5 | 4 | 9
    Past Use | 1 | 2 | 3
Alcohol abuse [Count of Participants; unit: Participants] — Population: Due to low baseline burden (<1%), 2 randomized subjects from each group were excluded from efficacy analysis.
  Participants | 0 | 1 | 1
Hypertension [Count of Participants; unit: Participants] — Population: Due to low baseline burden (<1%), 2 randomized subjects from each group were excluded from efficacy analysis.
  Participants | 4 | 4 | 8
Stroke [Count of Participants; unit: Participants] — Population: Due to low baseline burden (<1%), 2 randomized subjects from each group were excluded from efficacy analysis.
  Participants | 1 | 0 | 1
Coronary Artery Disease [Count of Participants; unit: Participants] — Population: Due to low baseline burden (<1%), 2 randomized subjects from each group were excluded from efficacy analysis.
  Participants | 0 | 2 | 2
Hyperlipidemia [Count of Participants; unit: Participants] — Population: Due to low baseline burden (<1%), 2 randomized subjects from each group were excluded from efficacy analysis.
  Participants | 3 | 4 | 7
Heart failure with reduced ejection fraction (HFrEF) [Count of Participants; unit: Participants] — Population: Due to low baseline burden (<1%), 2 randomized subjects from each group were excluded from efficacy analysis.
  Participants | 0 | 0 | 0
Heart failure with preserved ejection fraction (HFpEF) [Count of Participants; unit: Participants] — Population: Due to low baseline burden (<1%), 2 randomized subjects from each group were excluded from efficacy analysis.
  Participants | 0 | 0 | 0
Peripheral vascular disease (PVD) [Count of Participants; unit: Participants] — Population: Due to low baseline burden (<1%), 2 randomized subjects from each group were excluded from efficacy analysis.
  Participants | 0 | 0 | 0
COPD [Count of Participants; unit: Participants] — Population: Due to low baseline burden (<1%), 2 randomized subjects from each group were excluded from efficacy analysis.
  Participants | 0 | 0 | 0
Chronic renal failure/ kidney injury [Count of Participants; unit: Participants] — Population: Due to low baseline burden (<1%), 2 randomized subjects from each group were excluded from efficacy analysis.
  Participants | 0 | 0 | 0
Asthma [Count of Participants; unit: Participants] — Population: Due to low baseline burden (<1%), 2 randomized subjects from each group were excluded from efficacy analysis.
  Participants | 1 | 0 | 1
Diabetes mellitus [Count of Participants; unit: Participants] — Population: Due to low baseline burden (<1%), 2 randomized subjects from each group were excluded from efficacy analysis.
  Participants | 2 | 0 | 2
On chronic dialysis [Count of Participants; unit: Participants] — Population: Due to low baseline burden (<1%), 2 randomized subjects from each group were excluded from efficacy analysis.
  Participants | 0 | 0 | 0
Sleep disordered breathing [Count of Participants; unit: Participants] — Population: Due to low baseline burden (<1%), 2 randomized subjects from each group were excluded from efficacy analysis.
  Participants | 3 | 1 | 4
Previous open heart surgery [Count of Participants; unit: Participants] — Population: Due to low baseline burden (<1%), 2 randomized subjects from each group were excluded from efficacy analysis.
  Participants | 0 | 0 | 0
Coronary Artery Bypass Graft [Count of Participants; unit: Participants] — Population: Due to low baseline burden (<1%), 2 randomized subjects from each group were excluded from efficacy analysis.
  Participants | 0 | 0 | 0
Initial weight [Mean (Standard Deviation); unit: kilograms] — Population: Due to low baseline burden (<1%), 2 randomized subjects from each group were excluded from efficacy analysis.
  kilograms | 91.8 (12.2) | 102.8 (45.3) | 97.3 (32.1)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: Due to low baseline burden (<1%), 2 randomized subjects from each group were excluded from efficacy analysis.
  kg/m^2 | 30.9 (6.0) | 32.4 (11.1) | 31.6 (8.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in AF Burden
Description: Using mobile cardiac telemetry (MCT) to observe if AF burden is lower at 2 Weeks compared to Baseline in the active treatment group than the sham control group
Time Frame: 2 weeks
Population: We initially randomized 16 patients with paroxysmal AF. However, the DSMB decided that those with < 1% AF per week during the eligibility visit did not have sufficient AF burden to detect therapy effects. Therefore, all patients (2 in each group) with < 1% baseline AF burden were excluded from the analysis as screen failures. The remaining 12 included 8 men and 4 women with an average age of 60.9 ± 10.2 years
Measure: Mean (Inter-Quartile Range); unit: percentage of time in AF
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 6 | 6
percentage of time in AF | -0.4 [-7.9 to 4.22] | -2.4 [-14.1 to 16.6]

2. Secondary Outcome: Ventricular Rate Control
Description: Improved ventricular rate control during AF.
  AF-Free time was separated. Rate control during AF was categorized as the VR <=110 BPM stage.
Time Frame: 3 Months
Population: 1 patient who crossed over to the stimulation group did not have the 12-week visit
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 6 | 6
Participants
  Eligibility: AF-Free | 0 | 0
  Eligibility: VR ≤ 110 bpm | 4 | 4
  Eligibility: VR > 110 bpm | 2 | 2
  Week 1: AF-Free | 1 | 1
  Week 1: VR ≤ 110 bpm | 2 | 4
  Week 1: VR > 110 bpm | 3 | 1
  Week 2: AF-Free | 0 | 1
  Week 2: VR ≤ 110 bpm | 2 | 4
  Week 2: VR > 110 bpm | 4 | 1
  Week 3: AF-Free | 0 | 2
  Week 3: VR ≤ 110 bpm | 1 | 4
  Week 3: VR > 110 bpm | 5 | 0
  3 Months: number analyzed (Participants) | 6 | 5
  3 Months: AF-Free | 0 | 1
  3 Months: VR ≤ 110 bpm | 3 | 3
  3 Months: VR > 110 bpm | 3 | 1

3. Secondary Outcome: Average Skin Sympathetic Nerve Activity (SKNA)
Description: Reduction of SKNA taken from ME6000 (biomonitor) during Six Minute Walk test.
  SKNA is sympathetic nerve activity (SNA) recording from a skin-patch electrode used with the ME6000.
Time Frame: 3 months
Population: We initially randomized 16 patients with paroxysmal AF. However, the DSMB decided that those with < 1% AF per week during the eligibility visit did not have sufficient AF burden to detect therapy effects. Therefore, all patients (2 in each group) with < 1% baseline AF burden were excluded from the analysis as screen failures. The sham group was given the option to crossover to the experimental group after Week 3. One participant crossed over, therefore for month 3 data, N = 5.
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | Experimental Group | Control (Sham) Group
Number analyzed (Participants) | 6 | 6
microvolts
  Baseline - Lead 1 - At Rest | 0.93 (0.30) | 1.12 (0.85)
  Baseline - Lead 2 - At Rest | 0.89 (0.30) | 0.85 (0.11)
  Baseline - Lead 1 - Stress | 2.15 (0.76) | 1.65 (0.32)
  Baseline - Lead 2 - Stress | 1.98 (0.46) | 1.59 (0.45)
  Baseline - Lead 1 - Recovery | 1.45 (0.28) | 1.27 (0.39)
  Baseline - Lead 2 - Recovery | 1.23 (0.27) | 0.97 (0.26)
  Procedure - Lead 1 - At Rest | 1.31 (0.36) | 1.06 (0.29)
  Procedure - Lead 2 - At Rest | 1.69 (0.84) | 1.00 (0.30)
  Week 1 - Lead 1 - At Rest | 0.97 (0.52) | 0.95 (0.31)
  Week 1 - Lead 2 - At Rest | 0.88 (0.47) | 0.85 (0.26)
  Week 1 - Lead 1 - Stress | 2.12 (0.54) | 1.55 (0.20)
  Week 1 - Lead 2 - Stress | 1.92 (0.61) | 1.43 (0.28)
  Week 1 - Lead 1 - Recovery | 1.78 (1.47) | 1.13 (0.22)
  Week 1 - Lead 2 - Recovery | 1.08 (0.27) | 0.94 (0.17)
  Week 2 - Lead 1 - At Rest | 0.98 (0.53) | 0.89 (0.23)
  Week 2 - Lead 2 - At Rest | 0.88 (0.45) | 0.74 (0.22)
  Week 2 - Lead 1 - Stress | 2.16 (0.55) | 1.65 (0.35)
  Week 2 - Lead 2 - Stress | 1.95 (0.51) | 1.41 (0.21)
  Week 2 - Lead 1 - Recovery | 1.19 (0.27) | 1.15 (0.24)
  Week 2 - Lead 2 - Recovery | 0.93 (0.18) | 0.84 (0.13)
  Week 3 - Lead 1 - At Rest | 0.85 (0.27) | 1.05 (0.39)
  Week 3 - Lead 2 - At Rest | 0.74 (0.26) | 0.88 (0.33)
  Week 3 - Lead 1 - Stress | 2.26 (0.54) | 1.69 (0.44)
  Week 3 - Lead 2 - Stress | 2.11 (0.52) | 1.60 (0.37)
  Week 3 - Lead 1 - Recovery | 1.44 (0.35) | 1.40 (0.86)
  Week 3 - Lead 2 - Recovery | 1.14 (0.28) | 0.87 (0.19)
  Month 3 - Lead 1 - At Rest: number analyzed (Participants) | 6 | 5
  Month 3 - Lead 1 - At Rest | 1.04 (0.48) | 1.26 (0.64)
  Month 3 - Lead 2 - At Rest: number analyzed (Participants) | 6 | 5
  Month 3 - Lead 2 - At Rest | 0.93 (0.34) | 0.82 (0.19)
  Month 3 - Lead 1 - Stress: number analyzed (Participants) | 6 | 5
  Month 3 - Lead 1 - Stress | 2.20 (0.56) | 1.86 (0.62)
  Month 3 - Lead 2 - Stress: number analyzed (Participants) | 6 | 5
  Month 3 - Lead 2 - Stress | 2.00 (0.53) | 1.49 (0.33)
  Month 3 - Lead 1 - Recovery: number analyzed (Participants) | 6 | 5
  Month 3 - Lead 1 - Recovery | 1.42 (0.45) | 1.57 (0.14)
  Month 3 - Lead 2 - Recovery: number analyzed (Participants) | 6 | 5
  Month 3 - Lead 2 - Recovery | 1.10 (0.37) | 1.01 (0.13)

4. Secondary Outcome: Quality of Life - EQ-5D-5L
Description: Improvement of quality of life as measured by the EQ-5D-5L
Time Frame: 3 months
Population: EQ-5D-5L index scores range from -0.59 to 1, where 1 is the best possible health state. EQ-5D-5L health scores range from 5 (11111) to 25 (55555), where 5 is the best possible health state.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 6 | 6
score on a scale
  Baseline (total score) | 7.7 (4.6) | 6.3 (0.8)
  Week 3 (total score) | 7.2 (3.0) | 6.2 (0.8)
  Week 12 (total score) | 9.3 (5.9) | 6.0 (0.7)
  Baseline (index value) | 0.8 (0.4) | 0.9 (0.1)
  Week 3 (index value) | 0.8 (0.2) | 0.9 (0.0)
  Week 12 (index value) | 0.7 (0.5) | 0.9 (0.0)

5. Secondary Outcome: Quality of Life - AFEQT
Description: Improvement of quality of life as measured by the Atrial Fibrillation Effect on QualiTy-of-Life (AFEQT) Questionnaire. A score of 0 indicates the most severe symptoms or disability and a score of 100 indicates no limitation or disability. Thus, higher scores on the AFEQT instrument indicate better health status.
Time Frame: 3 months
Population: Overall or subscale scores range from 0-100.
  A score of 0 corresponds to complete disability (or responding "extremely" limited, difficult or bothersome to all questions answered), while a score of 100 corresponds to no disability (or responding "not at all" limited, difficult or bothersome to all questions answered).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 6 | 6
units on a scale
  Baseline AFEQT Global Score | 65.7 (29.8) | 49.7 (28.5)
  Week 3 AFEQT Global Score | 61.6 (28.4) | 63.1 (15.3)
  Week 12 AFEQT Global Score | 63.9 (29.9) | 71.7 (20.7)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for participants from Eligibility timepoint until Week 12/Month 3 MCT monitoring was completed.
Description: A crossover option was only given to those randomized to sham group initially, after the completion of the primary endpoint (Week 3 FU).
Groups:
- Control Group Crossed Over to Experimental: 1 sham participant chose to crossover and did not experience any adverse events to report.
Arm/Group | Experimental Group | Control Group | Control Group Crossed Over to Experimental
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/8 | 0/1
Other Adverse Events (participants affected / at risk) | 6/8 | 7/8 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Group (N=8) | Control Group (N=8) | Control Group Crossed Over to Experimental (N=1)
NA (elective left heart catheterization) (Cardiac disorders) | 1 | 0 | 0 — Underwent elective left heart catheterization (DES to RCA)
NA (elective left heart catheterization) (Cardiac disorders) | 1 | 0 | 0 — Underwent elective left heart catheterization (PCI to LAD)
Brief "Black Out" Periods (Cardiac disorders) | 1 | 0 | 0 — Hospitalization following a syncopal episode
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Group (N=8) | Control Group (N=8) | Control Group Crossed Over to Experimental (N=1)
NA (Skin Irritation) (Skin and subcutaneous tissue disorders) | 4 | 7 | 0 — Skin irritation from MCT patch electrode
NA (Bleeding) (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 — Bleeding from the insertion site
NA (Pain) (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 — Pain localized at lead site/stimulation point
NA (Goosebumps) (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 — Goosebumps during stimulation
NA (Hot Flashes) (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 — Hot flashes post-stimulation
NA (Skin Redness) (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Extremity weakness, swelling, and/or pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 — Neck, back, finger, leg joint pains
Allergic reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 — Allergic reaction to Tegaderm

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-19): https://cdn.clinicaltrials.gov/large-docs/41/NCT04529941/Prot_SAP_002.pdf
  • Informed Consent Form (2022-11-21): https://cdn.clinicaltrials.gov/large-docs/41/NCT04529941/ICF_001.pdf